CLINICAL TRIAL: NCT00573014
Title: Evaluating the Need for Magnetic Resonance Imaging of the Cervical Spine in Obtunded Trauma Patients
Brief Title: Cervical Spine Clearance in Obtunded Trauma Patients
Acronym: CSclearance
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB04-00110; IRB04-00110
Record Dates: First submitted 2007-12-10; First posted 2007-12-13 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Coma; Wounds and Injuries
Keywords: Obtunded blunt trauma patients
MeSH Terms: conditions — Coma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OBTP: Obtunded blunt trauma patients with normal CT C-spine
  Interventions: Other: Cervical Spine Clearance

INTERVENTIONS:
Other: Cervical Spine Clearance — All OBTPs with gross movement of all four extremities admitted to MetroHealth Medical Center who underwent a CT CS at MHMC between October 2006 and September 2008 will be included. Prospective data will be collected on these patients including age, gender, mechanism of injury, Glasgow Coma Scale (GCS) on admission, results of CT CS, GCS at the time of collar clearance, day of collar clearance, collar complications, date of reexamination, and results of reexamination. We will define an obtunded patient as a patient who was unable to reliably describe the presence or absence of CS symptoms in the opinion of the examining physician. Patients needed to have gross movement of all four extremities to be included in the study. We defined cervical collar complications as skin breakdown identified either by the skin care team during weekly rounds in the intensive care unit or by the treating physician at any time.

SUMMARY:
The optimal method of clearing the cervical spine in obtunded trauma patients is unclear. Computed tomography (CT) identifies most injuries but may miss ligamentous injuries. Magnetic resonance (MR) imaging has been widely used to exclude ligamentous injuries. We postulate that with the new generation of CT scanners, MR imaging is not needed to rule out significant injuries. Our protocol for clearing the cervical spine in obtunded trauma patients depends on CT alone. We are prospectively following these patients and performing a clinical examination when they are awake to show this is a safe approach.

DETAILED DESCRIPTION:
All OBTPs with gross movement of all four extremities admitted to MetroHealth Medical Center (MHMC), the regional Level I Trauma Center in Cleveland OH, who underwent a CT CS at MHMC between October 2006 and September 2008 will be included. Prospective data will be collected on these patients including age, gender, mechanism of injury, Glasgow Coma Scale (GCS) on admission, results of CT CS, GCS at the time of collar clearance, day of collar clearance, collar complications, date of reexamination, and results of reexamination. We will define an obtunded patient as a patient who was unable to reliably describe the presence or absence of CS symptoms in the opinion of the examining physician. Patients needed to have gross movement of all four extremities to be included in the study; if they did not, they were excluded. The presence or lack of sensory examination was not evaluated for the purposes of this study. We will define cervical collar complications as skin breakdown identified either by the skin care team during weekly rounds in the intensive care unit or by the treating physician at any time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will include all patients (including children) after blunt trauma in whom cervical spine injury has not been ruled out admitted to MetroHealth Medical Center from 10/1/2004-9/30/2006.

Exclusion Criteria:

* We are excluding patients with an obvious neurologic deficit attributable to the cervical spine.
* We are excluding patients with abnormalities of the cervical spine that are identified on either plain films or CT.
* We are also excluding those patients in whom the cervical spine can be cleared clinically due to normal mental status.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will include all patients (including children) after blunt trauma in whom cervical spine injury has not been ruled out admitted to MetroHealth Medical Center from 10/1/2004-9/30/2006. We are excluding patients with an obvious neurologic deficit attributable to the cervical spine. We are excluding patients with abnormalities of the cervical spine that are identified on either plain films or CT. We are also excluding those patients in whom the cervical spine can be cleared clinically due to normal mental status.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2008-07-01 (Actual); Study Completion 2008-09-30 (Actual)

PRIMARY OUTCOMES:
We postulate that with the new generation of CT scanners, MR imaging is not needed to rule out significant injuries. We hope to show that CT alone can be used to clear the cervical spine in obtunded trauma patients. | 2 years
  One hundred ninety-seven patients had their collars removed and CS cleared at a mean of 3.3 days. Removal of CS precautions in OBTPs with gross movement of all extremities is safe and efficacious if CT CS is negative for injury. Supplemental MRI CS is not needed in this patient population. Key Words: Magnetic resonance imaging, Computed tomography, Cervical

CONTACTS AND LOCATIONS:
Overall Officials: John J Como, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States